CLINICAL TRIAL: NCT06635356
Title: Evaluation of Sarcopenia in Patients Undergoing Knee Prosthesis
Brief Title: Knee Replacement and Sarcopenia
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Nida Lale, Assistant Doctor, Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Other Study IDs: IstanbulPMRTRH-kneerepsarc
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Sarcopenia; Knee Prosthesis; Knee Arthroplasty, Total
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- The frequency and change of sarcopenia in patients undergoing knee arthroplasty: Sarcopenia frequency and changes will be investigated in women and men between the ages of 50 and 75 who will undergo knee prosthesis surgery, with follow-ups to be performed before the operation, in the first month and in the third month after the operation.

SUMMARY:
The presence of sarcopenia in patients planned to undergo knee prosthesis and the effect of knee prosthesis on sarcopenia will be investigated

DETAILED DESCRIPTION:
Volunteer patients who will undergo knee replacement surgery in orthopedic clinics located in the Istanbul region and who meet the inclusion criteria will be recruited. A total of 31 volunteers will be included in the study.

First, all patients will be asked about their gender, age, height, weight, education, smoking, lifestyle, additional diseases, and treatments they have received. Then, a brief orthopedic evaluation will be performed on the patient. TANITA BIA analysis and grip strength measurement from the dominant hand will be performed on all patients before the operation, at 1 month and 3 months after the operation. Maximal voluntary grip strength will be measured with a hand dynamometer. Measurements will be made three times. For this measurement, the subject will be asked to hold a maximal voluntary grip for five seconds. There will be a ten-second rest period between the three tests. Measurements will be made with the JAMAR Plus+ (by Sammons Preston) hand dynamometry device. Before the test measurements, the patient will be shown how to use the device as an application. The highest of the three measured values will be taken. In addition, the calf circumference will be measured. While the patient is standing, the measurement will be made with a tape measure from the thickest point of the right and left calves without squeezing the skin. The same measurement will be repeated with the patient seated. At the same time, patients will be evaluated with walking speed test, sit-to-stand test, SARC-F, FRAIL Frailty Questionnaire, Mini Nutritional Assessment, EQ-5D General Quality of Life Scale, GLIM Test, Barthel Activities of Daily Living Index, CIRS Scale before the operation, 1st month and 3rd month after the operation.

When performing the walking speed test, the patient will be asked to walk as they normally do. A 4-meter or 3-meter walking speed test will be performed and a single test will be scored. Measurements will be made twice and the fastest will be evaluated.

In the sit-to-stand test, the person will be asked to try to get up without using their arms. If they cannot complete the test or can get up using their arms, the patient will receive 0 (zero) points. If they can get up using their arms, the repeated sit-to-stand test will be performed. In the repeated sit-to-stand test, the person will be asked to sit down and get up from a chair 5 times in a row without using their arms. Scoring will be between 0-4 depending on the time spent.

ELIGIBILITY:
Inclusion Criteria:

* Being between 50-75 years old
* Undergoing knee arthroplasty surgery
* Patients who agreed to participate in the study and gave written consent

Exclusion Criteria:

* Having a history of malignancy
* Being under 50 and over 75 years old
* Having one of the muscle/nerve diseases

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female or male patients between the ages of 50-75 who underwent knee arthroplasty surgery in orthopedic clinics in Istanbul
Sampling Method: Probability Sample
Enrollment: 31 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-04-03 (Estimated); Study Completion 2025-04-03 (Estimated)

PRIMARY OUTCOMES:
Calf circumference measurement | before surgery, 1st month after surgery, 3rd month after surgery
  Calf circumference is an anthropometric measurement that indicates fatfree muscle mass and has been considered by the World Health Organization (WHO) the most sensitive index for evaluating the decrease in muscle mass.
  While the patient is standing, the measurement will be taken with a tape measure from the thickest point of the right and left calves without squeezing the skin.
Handgrip strength | before surgery, 1st month after surgery, 3rd month after surgery
  Handgrip strength will be measured using a Jamar hand grip dynamometer (Model 5030J1, Sammons Preston Rolyan, Bolingbrook, Illinois, USA). Measurements will be taken 3 times in a sitting position with the elbow flexed to 90° and the wrist in neutral position. The measured maximal grip strength will be recorded as hand grip strength.
Skeletal muscle mass | before surgery, 1st month after surgery, 3rd month after surgery
  Skeletal muscle mass will be evaluated using a Tanita DC-360 multi-frequency body composition analysis device.
Body Mass Index (BMI) | before surgery, 1st month after surgery, 3rd month after surgery
  BMI will be calculated as weight (kg) divided by height2 (m2)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tanaka S, Kayamoto A, Terai C, Nojiri S, Fugane Y, Mori T, Nagaya M, Kako M, Iida H, Osawa Y, Takegami Y, Nishida Y. Preoperative Sarcopenia Severity and Clinical Outcomes after Total Hip Arthroplasty. Nutrients. 2024 Jun 29;16(13):2085. doi: 10.3390/nu16132085. PMID 38999833
- [Background] Tzartza CL, Karapalis N, Voulgaridou G, Zidrou C, Beletsiotis A, Chatziprodromidou IP, Giaginis C, Papadopoulou SK. Comparative Analysis on the Effect of Sarcopenia in Patients with Knee Osteoarthritis before and after Total Knee Arthroplasty. Diseases. 2023 Feb 22;11(1):36. doi: 10.3390/diseases11010036. PMID 36975585
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372